CLINICAL TRIAL: NCT05666089
Title: Effect of N-acetylcysteine Versus Calcium Hydroxide Used as an Intracanal Medicament on the Intensity of Postoperative Pain, Bacterial Load Reduction and Levels of MMP -9 in Periapical Fluids in Patients With Necrotic Pulp: A Randomized Clinical Trial
Brief Title: Effect of N-acetylcysteine Versus Calcium Hydroxide Used as an Intracanal Medicament on the Intensity of Postoperative Pain, Bacterial Load Reduction and Levels of MMP -9 in Periapical Fluids in Patients With Necrotic Pulp
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safwa Essam Mohammed Ahmed Abd el-glil, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: safwaendo91
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Intracanal Medication; N-acetylcystine; Calcium Hydroxide; Mediators
MeSH Terms: interventions — Acetylcysteine; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): intracanal medication of NAC paste
  Interventions: Drug: N-acetyl cysteine
- Calcium hydroxide (Active Comparator): intracanal medication of Ca(OH)2 paste
  Interventions: Drug: Calcium hydroxide

INTERVENTIONS:
Drug: N-acetyl cysteine — intracanal medication of NAC with concentration 1 gm/ml in the form of a paste
  Arms: N-acetylcysteine
Drug: Calcium hydroxide — intracanal medication of calcium hydroxide paste (metapaste)
  Arms: Calcium hydroxide

SUMMARY:
To compare the effect of N-acetylcysteine versus calcium hydroxide as intra canal medication on:

* Intensity of postoperative pain.
* Bacterial load reduction.
* levels of MMP -9 in Periapical Fluids.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition.
* Males & Females with

  * Mandibular single rooted permanent premolar teeth.
  * Absence of spontaneous pain.
  * Slight widening in the periodontal membrane space or with periapical radiolucency not exceeding 2*2 mm radiographically.
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent (Appendix I)

Exclusion Criteria:

1. Medically compromised patients.
2. Pregnant women
3. Patients undergoing previous endodontic treatment or analgesics and/or antibiotics have been administrated by the patient during the past 24 hours preoperatively.
4. Patients reporting bruxism or clenching.
5. Teeth that show association with acute periapical abscess and swelling.
6. Greater than grade I mobility or pocket depth greater than 5mm.
7. Non-restorable teeth or teeth that could not be adequately isolated with a rubber dam
8. Teeth with vital pulp.
9. Immature teeth.
10. Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 6 hours post-instrumentation.
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 12 hours post-instrumentation
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 24 hours post-instrumentation
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 48 hours post-instrumentation
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 6 hours post-obturation.
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 12 hours post-obturation
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 24 hours post-obturation
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)
Intensity of postoperative pain | 48 hours post-obturation
  Intensity of postoperative pain will be measured using numerical rating scale (NRS)

SECONDARY OUTCOMES:
Bacterial load reduction | Sample 1 (S1): after access preparation and pre-instrumentation.
  Bacterial counting using agar Culture technique
Bacterial load reduction | Sample 2 (S2): at the end of 1st visit post-instrumentation.
  Bacterial counting using agar Culture technique
Bacterial load reduction | Sample 3 (S3): after 2 weeks intracanal medicament placement (pre-obturation)
  Bacterial counting using agar Culture technique
Periapical MMP-9 level | at 1st visit post- instrumentation.
  using ELISA
Periapical MMP-9 level | after 2 weeks at 2nd visit (pre-obturation).
  using ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- FACULTY OF DENTISTRY-cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided